CLINICAL TRIAL: NCT04086927
Title: Unna Boot: a Technique to Decrease Preoperative Soft Tissue Swelling Following Ankle Fractures
Brief Title: Unna Boots for Ankle Fracture Swelling
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00092143
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients will not receive compression dressing
- Experimental Group (Experimental): Patients will receive compression dressing
  Interventions: Device: Unna Boot

INTERVENTIONS:
Device: Unna Boot — The unna boot is a zinc coated compression dressing
  Arms: Experimental Group

SUMMARY:
This study will evaluate the difference in soft tissue swelling prior to surgery and wound complications after surgery between unna boot application versus standard splint application. An unna boot is an extra zinc covered wrap around your leg followed by standard splint application (cotton dressing, plaster, then soft dressing). Prior to surgery the participant's swelling will be measured and compared to the standard splint application group. After surgery, the participant will be monitored for wound complications, pain, and range of motion.

DETAILED DESCRIPTION:
The purpose of this study is to compare preoperative swelling and frequency of wound complications in ankle fractures through standard splint and an unna boot compressive dressing with a splint. Quantitative and qualitative measurements will be analyzed to compare edema and wound complications. Secondary goals are to evaluate the quantitative differences in ankle range of motion and visual analogue scale (VAS) pain scores. The hypothesis of this proposed study is that there will be less soft tissue swelling and wound complications with the use of an unna boot when compared to the standard splint. The investigators also hypothesize that there will be improved ankle range of motion and visual analogue scale (VAS) pain scores with the use of an unna boot when compared to a standard splint. Participants will be randomized to either the standard splint or an unna boot and quantitative and qualitative measures will be collected. This data could change the practice for preoperative management of soft tissue swelling following ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

* acute ankle fracture

Exclusion Criteria:

* low energy ankle fracture
* open ankle fracture
* unwillingness to participate
* allergy to zinc
* revision surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Baseline swelling using Figure-8 Measurement | Baseline (Initial encounter)
  Physician uses tape measure to measure angles to determine swelling severity of ankle. This measurement is taken by making a figure eight pattern on the foot and ankle. The measurement is taken three times and then averaged to give the final total.
Mean swelling using Figure-8 Measurement | 6 weeks follow up visit
  Physician uses tape measure to measure angles to determine swelling severity of ankle. This measurement is taken by making a figure eight pattern on the foot and ankle. The measurement is taken three times and then averaged to give the final total.
Mean pain scores on visual analogue scale at initial encounter | Baseline (initial encounter)
  patients report a pain score of 1-10. 1 being the lowest and 10 being the highest
Mean pain scores on visual analogue scale at 6 week follow up visit | 6 weeks follow up visit
  patients report a pain score of 1-10. 1 being the lowest and 10 being the highest

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Gross, M.D., Principal Investigator — Orthopaedic Surgeon